CLINICAL TRIAL: NCT06502275
Title: Effects of the Tailored Frailty Prevention Program With Exercise and Nutrition Management to Improve Physical Performance and Health Status in Older Patients With Colorectal Cancer
Brief Title: Nutrition and Exercise Program for Elderly Colorectal Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ching-Ching Su, Assistant Professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202300957B0C601
Record Dates: First submitted 2024-07-08; First posted 2024-07-16 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
Keywords: Older; Colorectal cancer; Frailty; mobile health; Physical activity; nutrition
MeSH Terms: conditions — Colorectal Neoplasms; Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrition combined with exercise group (Experimental): Provide mobile health interventions that combine nutrition and exercise
  Interventions: Behavioral: Mobile Health Management Frailty Care Program
- routine care group (No Intervention): Provide routine care

INTERVENTIONS:
Behavioral: Mobile Health Management Frailty Care Program — Through the "LINE" communication software, participants are provided with exercise and nutrition information three times a week, with a total of 36 messages. As well as 6 podcasts of health information and 6 sports videos in total. At weeks 2, 4, and 6, researchers scheduled 5- to 10-minute telephone consultations. Participants can receive guidance through telephone consultations and carry a Xiaomi sports band wearable device to monitor their exercise.
  Arms: Nutrition combined with exercise group

SUMMARY:
The goal of this interventional study is to evaluate the effect of mobile health intervention on frailty, physical fitness, physical activity, and nutritional status of elderly patients with colorectal cancer. The main questions it aim to answer are: 1. Does the mobile health intervention reduce frailty in elderly colorectal cancer patients compared to standard care? 2. Does the mobile health intervention improve physical fitness, physical activity, and nutritional status in elderly colorectal cancer patients compared to standard care? Participants will receive the Mobile Health Management Frailty Care Program.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colorectal cancer confirmed by a physician.
* Aged 60 and above.
* Have communication skills, able to read and write or converse in Mandarin and Taiwanese.
* Clear consciousness and no mental or cognitive impairment.
* Physical activities are accessible.
* Those who have a smartphone and have experience using smartphones.

Exclusion Criteria:

* People who have difficulty walking or standing.
* The wrist is not suitable for those wearing sports bracelets.
* People in infectious or protective isolation.
* Those who live alone or in institutions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Frailty | Pre-test, sixth week after intervention, 13th week after intervention
  Assessing frailty status using the G8 geriatric screening tool. Scores range from 0 to 17, with 0 indicating severe impairment and 17 indicating no impairment. The lower the score, the more frail it is.
Physical Activity | Pre-test, sixth week after intervention, 13th week after intervention
  Assess physical activity with the International Physical Activity Questionnaire-Short Form. The IPAQ-SF evaluates the number of days and time spent performing MVPA, walking, and sitting in bouts of at least 10 min over the previous 7 days. The summary score is expressed in PA metabolic equivalent of task (MET)-min per day or week.
Nutritional Status | Pre-test, sixth week after intervention, 13th week after intervention
  Assess nutritional status with Mini Nutritional Assessment-Short Form. The total score is 0-14 points. A score of 12 or more indicates a low risk of malnutrition. A score of 8-11 indicates a potential risk of malnutrition. A score less than 7 indicates a high risk of malnutrition.

SECONDARY OUTCOMES:
health-related quality of life | Pre-test, sixth week after intervention, 13th week after intervention
  Assessing quality of life using Taiwan Chinese version of European Organization for Research and Treatment of Cancer questionnaires. For all scales, item scores are summed and linearly transformed into a scale ranging from 0 to 100. Higher scores on the functioning scales indicate higher levels of functioning
Depression | Pre-test, sixth week after intervention, 13th week after intervention
  Assessing depression level using the Geriatric Depression Scale Short Form. The higher the score, the higher the degree of depression. 0-4 indicates normal, 5-10 indicates slight tendency to depression, and 10 or more indicates symptoms of depression.
body mass index | Pre-test, sixth week after intervention, 13th week after intervention
  Body mass index is calculated by dividing weight (kg) by height (meters) squared. The normal range is 18.5 ≦ BMI < 24. Less than 18.5 represents underweight; 24 ≦ BMI <27 represents overweight; 27 ≦ BM I<30 represents mild obesity; 30 ≦ BMI <35 represents moderate obesity; BMI ≧35 represents severe obesity.
hand grip strength | Pre-test, sixth week after intervention, 13th week after intervention
  Hand grip strength (in kilograms) was measured using a digital hand dynamometer (EH101; Camry, Guangdong Province, China). The grip strength of the dominant hand was assessed three times, and the maximal value was considered for analysis. The definition of normal GS according to European Working Group on Sarcopenia in Older People (EWGSOP) was ≥ 30kg in the male and ≥ 20 kg in the female. Weak GS was defined as GS < 30 kg in the male and GS < 20 kg in the female.
walking speed | Pre-test, sixth week after intervention, 13th week after intervention
  Walking speed was measured with a 4-meter walking evaluation with a static start. The 4-m gait speed was assessed to the nearest 0.01 s using a stopwatch. Participants were instructed to walk at their comfortable speed. Walking distance exceeded the required four meters to prevent participants from slowing down before reaching the 4-m line. The fastest time of two trials was used for analyses and gait speed was expressed in m/s. The 0.8 m/s cut-point was used to represent a slow walking speed.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ching Su, PhD, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No